CLINICAL TRIAL: NCT00748540
Title: Clinical Trial of the Vibrant Soundbridge as a Treatment for Conductive and Mixed Hearing Losses, Using Direct Round Window Cochlear Stimulation.
Brief Title: Safety and Efficacy of the Vibrant Soundbridge (VSB) for Mixed and Conductive Hearing Losses
Acronym: VSBRW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Med-El Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G060227
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Results first posted 2018-07-31 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Hearing Loss
Keywords: sensorineural hearing loss; conductive hearing loss; mixed hearing loss
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sensorineural; Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Implanted (Experimental): Implanted with Vibrant Soundbridge
  Interventions: Device: Vibrant Soundbridge

INTERVENTIONS:
Device: Vibrant Soundbridge — Mixed and conductive hearing loss using round window stimulation
  Other Names: VSB; VSB RW; RW VSB; Round Window Stimulation

SUMMARY:
The purpose of this investigation is to collect feasibility data to assess the safety and efficacy of the Vibrant Soundbridge (VSB), a medical device designed to provide benefit in aided hearing thresholds, speech perception and sound quality to certain individuals with hearing loss with minimal changes in residual hearing. The VSB is currently indicated for adults with moderate-to-severe sensorineural hearing loss. Under the present investigation, adults with conductive and mixed hearing losses who are not successful users of traditional amplification will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 years of age or older at time of implantation
* English as the primary language
* Appropriate motivation and expectation levels
* Geographically and physically able to return to the investigational center for scheduled evaluations and follow-up appointments.
* At least a 28-day unsuccessful hearing aid trial (within the past 24 months prior to enrolment).
* Persons who after being informed that a different hearing aid than the one they currently have may provide improved hearing, still request an implant.
* Ability to undergo general anesthesia
* Audiological tests suggest either a conductive or mixed hearing loss. The non-implanted ear may fall outside these criteria; however, threshold levels may not be worse than severe sloping to profound.
* Conductive Hearing Loss
* Pure-tone bone-conduction threshold levels in the ear to be implanted shall fall at or within the levels stated below. There should be an air-bone gap of 15 dB HL or more at three or more of the frequencies 500, 1000, 1500, 2000, 3000, and 4000 Hz. Pure-tone air-conduction levels should indicate the presence of at least a moderate hearing loss of at least 41 dB HL. Air conduction levels are not limited on the upper end.
* Upper Limits of Bone Conduction Thresholds for Conductive Hearing Loss Frequency (kHz) 0.5 1.0 1.5 2.0 3.0 4.0 Bone Conduction upper limit (dBHL) <25 <25 <25 <25 <25 <25
* Mixed Hearing Loss
* Pure-tone bone conduction threshold levels in the ear to be implanted shall fall at or within the levels stated below. There should be an air-bone gap of 15 dB HL or more at three or more of the frequencies 500, 1000, 1500, 2000, 3000, and 4000 Hz. Bone conduction thresholds at least three of the frequencies should be 26 dB or greater. Pure-tone air-conduction thresholds should be, on average, at least moderately impaired of 41 dB or greater. Air-conduction levels are not limited on the upper end.
* Lower and Upper Limits of Bone Conduction Thresholds for Mixed Hearing Loss Frequency (kHz) 0.5 1.0 1.5 2.0 3.0 4.0 Bone Conduction lower limit (dBHL) 0 0 0 0 0 0 Bone Conduction upper limit (dBHL) 45 50 55 65 65 65
* Good potential for aided speech recognition as indicated by a pre-operative monosyllabic word score of > 30% in the ear to be implanted as measured under headphones at 40 dB SL or at MCL
* Hearing aid trial with appropriately fitted hearing aids of at least 28 days duration within the past 24 months, unless the subject is unable to wear hearing aids for medical reasons
* Most recent audiometric data, if available, judged to be of good test-retest reliability.

Exclusion Criteria:

* Hearing loss of purely sensorineural origin
* Retrocochlear or central auditory disorders
* Active middle ear infection
* Tympanic membrane perforation, ears with previously reconstructed tympanic membranes may be included
* Bone-conduction thresholds in the ear to be implanted that have demonstrated a recent fluctuation at two or more frequencies of 15 dB in either direction in the last 6 months, as demonstrated by serial audiograms.
* History of post-adolescent, inner-ear disorders, such as vertigo or labyrinthitis
* Chronic or non-revisable vestibular or balance disorders
* Middle ear infections not responsive to medical treatment
* Skin or scalp conditions that may preclude attachment of the Audio Processor or that may interfere with the use of the Audio Processor
* Chronic pain in or around the head
* Current or previous use of an active hearing implant in either ear.
* Any known physical, psychological, or emotional disorder that may interfere with the completion of scheduled follow-up evaluations
* Developmental delays or organic brain dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Foyt, MD, Principal Investigator — Capital Region Ear Institute; Jose Fayad, MD, Principal Investigator — House Ear Institute; Jennifer Maw, MD, Principal Investigator — Jennifer Maw, MD; Robert Cullen, MD, Principal Investigator — Midwest Ear Institute; Douglas Chen, MD, Principal Investigator — Pittsburgh Ear Associates; Jack Wazen, MD, Principal Investigator — Silverstein Institute; Hinrich Staecker, MD, PhD, Principal Investigator — University of Kansas Medical Center; Fred Telischi, MD, Principal Investigator — University of Miami; Craig Buchman, MD, Principal Investigator — University of North Carolina Hospital; Peter Roland, MD, Principal Investigator — University of Texas Southwestern Medical Center; Richard Wiet, MD, Principal Investigator — Ear Institute of Chicago
Locations (11):
- United States (11):
  - House Ear Institute, Los Angeles, California
  - Jennifer Maw, MD, San Jose, California
  - University of Miami Ear Institute, Miami, Florida
  - Silverstein Institute, Sarasota, Florida
  - Ear Institute of Chicago, Hinsdale, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Midwest Ear Institute, Kansas City, Missouri
  - Capitol Region Ear Institute, Slingerlands, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - Pittsburgh Ear Associates, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Background] Colletti V, Soli SD, Carner M, Colletti L. Treatment of mixed hearing losses via implantation of a vibratory transducer on the round window. Int J Audiol. 2006 Oct;45(10):600-8. doi: 10.1080/14992020600840903. PMID 17062502
- [Background] Kiefer J, Arnold W, Staudenmaier R. Round window stimulation with an implantable hearing aid (Soundbridge) combined with autogenous reconstruction of the auricle - a new approach. ORL J Otorhinolaryngol Relat Spec. 2006;68(6):378-85. doi: 10.1159/000095282. Epub 2006 Oct 26. PMID 17065833

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Implanted
Started | 50
Completed | 49
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Implanted
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 47
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 46 [18 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Speech Perception in Quiet (Monosyllables) in Patients Implanted With Vibrant Soundbridge
Description: Percent correct on words in quiet at the preoperative interval compared to 6 month post operative interval.
Time Frame: 6 months post initial activation
Measure: Mean (Standard Deviation); unit: percentage of words correct
Arm/Group | Implanted
Number analyzed (Participants) | 49
percentage of words correct | 94.12 (6.25)

2. Secondary Outcome: Functional Gain Compared to Preoperative Unaided Condition in Patients Implanted With Vibrant Soundbridge.
Description: Auditory thresholds in the soundfield at the preoperative interval compared to the 6 month postoperative interval.
Time Frame: 6 months post initial activation
Measure: Count of Participants; unit: Participants
Arm/Group | Implanted
Number analyzed (Participants) | 49
Participants
  Improved | 44
  Worsened | 0
  No change | 5

3. Secondary Outcome: Speech Perception in Noise (HINT Sentences) in Patients Implanted With Vibrant Soundbridge.
Description: Signal to Noise Ratio for sentences at the preoperative interval compared to the 6 month interval.
Time Frame: 6 months post initial activation
Population: 3 subjects did not completed this testing due to limitations of the equipment used.
Measure: Mean (Standard Deviation); unit: Signal to Noise Ratio
Arm/Group | Implanted
Number analyzed (Participants) | 46
Signal to Noise Ratio | 0.24 (3.97)

4. Secondary Outcome: Residual Hearing in Patients Implanted With Vibrant Soundbridge
Description: Unaided hearing thresholds measured at the 10 month interval compared to the preoperative interval in order to assess any changes
Time Frame: 10 months post initial activation
Measure: Count of Participants; unit: Participants
Arm/Group | Implanted
Number analyzed (Participants) | 50
Participants
  Maintained residual hearing | 48
  Decreased residual hearing | 2

ADVERSE EVENTS:
Arm/Group | Implanted
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 2/50
Other Adverse Events (participants affected / at risk) | 17/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implanted (N=50)
Staph infection following revision surgery (Ear and labyrinth disorders) | 1 (1)
Device removal due to tuberculosis infection (Ear and labyrinth disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implanted (N=50)
Conductor link exposure (Ear and labyrinth disorders) | 5 (7)
FMT off the round window (Ear and labyrinth disorders) | 7 (7)
Electromagnetic interference (Ear and labyrinth disorders) | 5 (6)
Defective audio processor (Ear and labyrinth disorders) | 4 (4)
Recurrence of cholesteoma (Ear and labyrinth disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less